CLINICAL TRIAL: NCT04222777
Title: Analysis of Cervical Motion During Flexion and Extension Cinematographic Recordings in Asymptomatic Elderly
Brief Title: Cervical Spine Motion in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NL70381.096.19
Record Dates: First submitted 2019-10-29; First posted 2020-01-10 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Cervical Spine Degeneration; Movement, Abnormal; Aging
Keywords: Cervical Motion; Physiological movement; Cervical spine; Segmental Rage of Motion; Elderly; Lower Cervical Spine; Fundamental Research; Cinematographic recordings
MeSH Terms: conditions — Dyskinesias

STUDY DESIGN:
Intervention Model Description: Fundamental research. Cinemathographic recordings will be made in healthy volunteers to determine physiological range of motion in the cervical spine. No health outcome of the intervention will be assessed.
Masking Description: Not applicable. All participants are healthy volunteers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Heatlhy volunteers. (Other): Healthy volunteers will undergo two cinematographic recordings of the cervical spine
  Interventions: Diagnostic Test: Cinematographic Recording

INTERVENTIONS:
Diagnostic Test: Cinematographic Recording — A cinematographic recording during the second half of extension of the cervical spine will be made during 16 seconds at two timepoints with an interval of two weeks.

SUMMARY:
Rationale:

Physiological motion of the cervical spine is a subject of interest for medical specialists. Segmental range of motion (sROM) has been most commonly used to define motion but inter- and intra-variability is large. Therefore, a sequence of segmental contributions in the lower cervical spine during the second half of extension has been defined in healthy participants (uniform in 80-90%). The mean age of these participants was 23 years. Since cervical degenerative disc disease (CDDD) occurs more often in elderly patients, it is of paramount importance to study whether this sequence remains present during aging, regardless of losing 0.11 degrees of sROM each year.

Objective:

To investigate if the normal sequence of segmental contributions in the lower cervical spine during the second half of extension (C4-C5 followed by C5-C6, and then C6- C7) is also present in asymptomatic participants between 55 and 70 years of age by using cinematographic recordings.

Study design:

Fundamental research

Study population:

Eleven asymptomatic participants between 55 and 70 years of age, without a medical history of neck problems, with a score of 4 or less on the Neck Disability Index (NDI), and without severe degenerative changes based on a score of 3 or less on the radiological Kellgrens' classification.

Intervention:

Two flexion and extension cinematographic recordings of the cervical spine with a two-week interval between recordings.

Main study parameters/endpoints:

Primary endpoint: Defining the cervical spines' physiological motion pattern by analysing the normal sequence of segmental contributions in the lower cervical spine (C4-C5 followed by C5-C6, and then C6-C7) during the second halfof extension in asymptomatic participants between 55 and 70 years of age.

Secondary endpoint: Determine sROM of C4-C5, C5-C6, and C6-C7 by analysing the flexion and extension cinematographic recordings in asymptomatic participants between 55 and 70 years of age.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Participants receive cinematographic recordings twice. There will be no follow-up.

DETAILED DESCRIPTION:
INTRODUCTION AND RATIONALE Physiological motion of the cervical spine is a subject of interest for medical specialists. Although the term 'physiological motion' is commonly used, a proper definition has been lacking for a long time. Segmental range of motion (sROM, e.g. the amount of sagittal rotation in a segment between maximal flexion and maximal extension position of the entire cervical spine) is most commonly used to study motion. SROMs, however, suffer from large intra- and interindividual variability. Therefore, in the lower cervical spine, Boselie et al have recently described a consistent sequence of segmental contribution in sagittal rotation during flexion and extension in 20 healthy participants. This was based on historic reports. The mean age of the healthy participants was 23 years (SD 2.65, range 18-55 years). They showed that the sequence of segmental contributions in the lower cervical spine during the second half of extension of the entire cervical spine and head was uniform in 80-90% of the healthy participants. The sequence of segmental contributions was C4-C5 followed by C5-C6, and then C6-C7. Also, they described a group of single level cervical degenerative disc disease (CDDD) patients in which this sequence was present in only one patient (10%). This is the first method described which can reliably differentiate between normal or abnormal movement of the cervical spine in an individual subject. CDDD is degeneration of a cervical intervertebral disc and/or the adjoining vertebral bodies leading to cervical radiculopathy and/or myelopathy. CDDD occurs more often in elderly patients (> 50 years of age) and due to aging of the population this will become a larger problem in the future. Age has been shown to be associated with a 0.11 degree decrease of sROM per year, independent of degeneration. Given that there are five levels in the subaxial cervical spine, there is an associated five degrees decrease in motion of the total subaxial cervical spine for every 10 years of ageing. It remains unclear whether the normal sequence of segmental contributions in the lower cervical spine is also present in asymptomatic elderly. By confirming the normal sequence in this group, this can be used to determine abnormal motion in elderly patients suffering from CDDD. The intention is to use this in future research in patients with cervical myelopathy or radiculopathy undergoing surgery to compare the outcomes of different types of surgery (e.g. cervical arthroplasty or anterior cervical discectomy with fusion) and to compare the influence of the type of surgery on normal motion.

2. OBJECTIVES Primary Objective: To investigate whether the normal sequence of segmental contributions in the lower cervical spine during the second half of extension (C4-C5 followed by C5-C6, and then C6-C7), which is present in young asymptomatic controls, is similar in asymptomatic participants between 55 and 70 years of age by using cinematographic recordings.

Secondary objective: To determine sROM of C4-C5, C5-C6, and C6-C7 by analysing the flexion and extension cinematographic recordings in asymptomatic participants between 55 and 70 years of age.

3. STUDY DESIGN This is a fundamental research project in which asymptomatic elderly participants without neck pain or severe degenerative changes will be included. Participants will be recruited at Zuyd Hogeschool Sittard/Heerlen and Zuyderland Medical Center Sittard- Geleen/Heerlen by using posters notifying about the study. They can contact the researcher by email, who will inform them verbally and in writing. Informed consent will be signed if they meet the in- and exclusion criteria and if they are willing to participate. Flexion and extension of the cervical spine has been analysed through sagittal cinematographic recordings before. This was done in two groups with ten healthy participants in each group, from which an adequate analysis could be performed. Taking a possible loss to follow up of 10% into account, our study population will consist of 11 participants. No interim analysis will be performed. Each participant receives flexion and extension cinematographic recording twice to determine reproducibility and consistency of sequence between the two time points (T1 and T2). Recordings will be performed with an interval of two weeks, resulting in 22 cinematographic recordings. Inclusion is expected to take approximately three months. Possible participants have to complete the Neck Disability Index (NDI), participants scoring above 4/50 points will be excluded (which means they would be no longer be classified as 'no disability due to neck problems'). A lateral X-ray of the cervical spine will be made, which will be scored using Kellgrens' classification by two neurosurgeons to avoid inclusion of participants with severe degenerative changes. Participants with a Kellgren score (KS) of four will be excluded. A KS score of four indicates severe degenerative changes such as severe narrowing of the disc space, severe sclerosis of the vertebral plates, or multiple large osteophytes. Participants with KS between zero and three will be included, indicating no, minimal, or moderate degenerative changes.

4. STUDY POPULATION Population (base) Male and female participants between 55 and 70 years of age, without a history of neck complaints, an NDI score of 4 or less and a KS of 3 or less will be included. Participants will be recruited using posters in Zuyd Hogeschool Sittard/Heerlen and Zuyderland Medical Center Sittard- Geleen/Heerlen.

Sample size calculation Sample size calculation is based on previous articles using the same method of cinematographic recordings to analyse motion of the cervical spine. Our study population will consist of 11 participants, assuming a possible loss to follow-up of 10%. Flexion and extension cinematographic recordings are acquired twice for each participant with an interval of two weeks in order to determine reproducibility and consistency of sequence of motion between two time points (T1 and T2). If there is no loss to follow-up and all cinematographic recordings are of good quality in the first 10 participants, the study will be ended.

5. TREATMENT OF SUBJECTS 5.1 Investigational product/treatment Cinematographic recordings during flexion and extension of the cervical spine in asymptomatic elderly participants.

5.2 Use of co-intervention Not applicable.

5.3 Name and description of investigational product Not applicable.

5.4 Summary of findings from non-clinical studies Not applicable.

5.5 Summary of findings from clinical studies

Initially, a method was developed to determine the ROM in the sagittal plane of the cervical spine using a fluoroscopy video of flexion-extension movement. The total ROM (tROM) and the sROM in 10 healthy participants (19-22 years) was investigated. The tROM for anteflexion is 118.1 degrees and 114.3 degrees for retroflexion. Several new and very important insights have been published in this study. The maximum sROM is not necessarily reflected comparing the position of the vertebra in full flexion to its position in full extension. Moreover, sROM differs depending on execution of the motion from flexion to extension or the other way around and sROM can differ with time. A difference in excess of five degrees for the same segment in the same individual can be recorded. The cadence of movement in the cervical spine was also described. During flexion and extension, motion of the cervical vertebrae follows a general pattern which is complex and counter- intuitive. They conclude that tROM and sROM are unsuitable to be used as a parameter of cervical spine mobility.

A review that systematically addressed contemporary knowledge about the mechanical behaviour of cervical vertebrae and soft-tissue of the cervical spine, under conditions that result in minor of major injuries. The results are collected from multiple studies that have measured sROM of individual joints of the cervical spine. It is emphasised that, even under normal conditions, sROM is not consistent either in time or according to the direction of motion.

sROM and KS with flexion/ extension radiographs were assessed and the relation to clinical variables in 195 patients was determined (age 15-93 years, 62 males and 133 females). Interobserver reliabilities for assessing KS (intraclass correlation coefficient 0.81) and sROM (intraclass correlation coefficient 0.72) were good to excellent. Age had a significant negative association with sROM at C2-C3, C3-C4, C4-C5, and C5-C6, amounting to a total of five degrees decrease in subaxial cervical ROM every 10 years. KS at the level of interest had a significant negative association with sROM at C2-C3, C3-C4, C4- C5, C5-C6, and C6-C7. KS at the inferior segment had a significant positive association with sROM at C2-C3, C3-C4, and C4-C5. For every point increase in KS at a given level, there was an associated 1.2 degrees decrease in sROM at that level, and 0.8 degrees increase in sROM at the level above. Gender had a significant association with sROM only at C2-C3.

A non-invasive infrared system Polaris was used to quantify the 3D tROM of the cervical spine in 140 asymptomatic volunteers (age 20-93 years, 70 males and 70 females). The standard error of measurement for the maximum tROM in 3D space planes was 5%. Gender had no significant influence on the 3D cervical tROM. Age had a significant influence on all main movements showing 0.55 - 0.79 degrees magnitude decrease per decade per segment.

Later, an automatic fast and precise method for tracking cervical vertebrae in fluoroscopy videos of flexion- extension movement of the cervical spine was developed. The method relies only on a rough selection of template areas of each vertebra in a single frame of the video sequence, no contours need to be extracted and no vertebra segmentation is required. Tracking is done with a normalized gradient field, using only the gradient orientations as features. Results show that the algorithm is robust and able to track the vertebrae accurately, even if they are partially occluded or if a disc prosthesis is present.

A clear definition of the normal sequence of segmental contributions in the cervical spine using extension cinematographic recordings (ECRs) was defined. They analysed healthy participants (n=20) and patients with CDDD (n=10). ECRs were more consistent than flexion cinematographic recordings (FCRs) and were therefore used to define "normal" motion. A consistent sequence of contribution of sagittal rotation of the three lower cervical motion segments C4-C7 was especially identified in the last phase of extension in healthy participants. The first peak was found for C4- C5, followed by C5-C6 and finally in C6- C7. Sensitivity, specificity, and reliability were calculated. Reliability of scoring as normal or abnormal is high (Fleiss kappa of 0.80-0.84, range of 95% CI: 0.66- 0.98). Sensitivity and specificity are also high, with an average sensitivity of 90% (range of 95% CI: 78.4 - 99.8%), nd an average specificity of 85% (range of 95% CI: 72.9 - 96.4%). This is the first described method which can reliably differentiate between normal or abnormal movement of the cervical spine in an individual subject.5.6 Summary of known and potential risks and benefits Flexion- and extension cinematographic recordings are made using the Philips Allura Xper FD20 X-ray system. Radiation dose per cinematographic recording, determined by radiation experts, will be around 0.084 mSv. Participants will perform cinematographic recordings twice, resulting in a total radiation dose of 0.168 mSv. Moreover, before definitive inclusion in the study a lateral X-ray of the cervical spine will be performed to determine eligibility resulting in a radiation dose of 0.0096 mSv. Average radiation dose per participant will therefore be 0.1776 mSv. This amount of radiation can be categorized in category IIa using the Neurocritical Care Society (NCS) guidelines about risks of radiation dosage (0.1 to 1 mSv) 11. This category includes moderate risk which can be justified if there is a potential health benefit for future patients.

6. METHODS 6.1 Study parameters/endpoints

6.1.1 Main study parameter/endpoint To investigate whether the normal sequence of segmental contributions in the lower cervical spine during the second half of extension (C4-C5 followed by C5-C6, and then C6-C7), which is present in young asymptomatic controls, is similar in asymptomatic participants between 55 and 70 years of age by using cinematographic recordings. Recordings will be made at two occasions, with an interval of two weeks. These will then be analysed within one year.

6.1.2 Secondary study parameters/endpoints (if applicable) Analysing sROM of C4-C5, C5-C6 and C6-C7 by analysing the flexion and extension cinematographic recordings in asymptomatic participants between 55 and 70 years of age. Recordings will be made at two occasions, with an interval of two weeks. These will then be analysed within one year.

6.2 Randomisation, blinding and treatment allocation Not applicable.

6.3 Study procedures This study does not use invasive procedures, but is not regular care.

Investigations before inclusion in the study:

Lateral X-ray of the cervical spine to determine Kellgrens' classification. The KS will be determined by two neurosurgeons and is a scoring method to determine severity of degenerative disc disease, using five gradations :

Grade 0: absence of degeneration in the disc. Grade 1: minimal anterior osteophytosis. Grade 2: definite anterior osteophytosis, possible narrowing of the disc space, some sclerosis of the vertebral plates.

Grade 3: moderate narrowing of the disc space, sclerosis of the vertebral plates, osteophytosis.

Grade 4: severe narrowing of the disc space, severe sclerosis of the vertebral plates, multiple large osteophytes.

Questionnaire the NDI:

The NDI is a modification of the Oswestry Low Back Pain Disability Index. It is a patient- completed, condition-specific functional status questionnaire with 10 items including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation. Each section is scored on a 0 to 5 rating scale, in which zero means 'No pain' and 5 means 'Worst imaginable pain'. Al the points can be summed to a total score. The test can be interpreted as a raw score, with a maximum score of 50, or as a percentage. 0 points or 0% means: no activity limitations, 50 points or 100% means complete activity limitation.

Investigations during the study:

- Cinematographic recordings: participants are seated on a crutch, adjustable in height, with their neck, shoulders and head free. Before recordings are made, participants will be taught to perform the prescribed flexion and extension movement on about 16 seconds using a metronome. Participants are placed on the crutch with their shoulder's perpendicular to the image intensifier to obtain sagittal images from the occiput till C7. As soon as the recording is started, the participant is instructed to move his head in the sagittal plane from maximal ex- tension to maximal flexion, without moving the upper part of the body. It is important that the participants shoulders are kept as low as possible while making the recordings to ensure that all the cervical vertebrae are visible. The movement of the cervical spine should be as fluent as possible to prevent for sudden large rotations and translations between consecutive frames. The cinematographic recordings will be made twice with an interval of two weeks using the Philips Alura Xper FD20 X- ray system. To stay below the limit of 1 mSv per participant, the 0.9 mm Cu + 1 mm Al filter will be used for the entire study. The Alura Xper automatically selects correct tube voltage, with an expected maximum around 70-80 kV for cervical cinematographic recordings.

6.4 Withdrawal of individual subjects Participants can cease study participation at any time for any reason if they wish to do so, without any consequences. If participants leave the study before the second recording, only the first recording will be included and analysed.

Researchers cannot decide to withdraw participants from the study, unless participants do not respond to calls before the first cinematographic recording is made.

6.5 Replacement of individual subjects after withdrawal If a participant withdraws before the first cinematographic recording is made, researchers are allowed to replace this participant.cal cinematographic recordings.

6.6 Follow-up of subjects withdrawn from treatment Participants who withdraw from the study will not be actively recalled.

6.7 Premature termination of the study Interim analysis will not be performed, so there will be no reason to terminate the study prematurely.

7. SAFETY REPORTING 7.1 Temporary halt for reasons of subject safety In accordance to section 10, subsection 4, of the WMO, the investigator will suspend the study if there is sufficient ground that continuation of the study will jeopardise subject health or safety. The sponsor will notify the accredited METC without undue delay of a temporary halt including the reason for such an action. The study will be suspended pending a further positive decision by the accredited METC. The investigator will take care that all subjects are kept informed.

7.2 AEs, SAEs and SUSARs 7.2.1 Adverse events (AEs) Adverse events are defined as any undesirable experience occurring to a participant during the study, whether or not considered related to experimental intervention. All adverse events reported spontaneously by the participant or observed by the investigator or his staff will be recorded.

7.2.2 Serious adverse events (SAEs) A serious adverse event is any untoward medical occurrence or effect that results in: Death.

Is life threatening (at the time of event). Requires hospitalization or prolongation of existing inpatients' hospitalization. Results in persistent or significant disability or incapacity.

Is a congenital anomaly or birth defect. Any other important medical event that did not result in any of the outcomes listed above due to medical or surgical intervention but could have been based upon appropriate judgement by the investigator. An elective hospital admission will not be considered as a serious adverse event. The investigator will report all SAEs to the sponsor without undue delay of obtaining knowledge of the events. Sponsor will report these SAEs through the web portal ToetsingOnline to the accredited METC that approved the protocol, within 7 days for SAEs that result in death or life- threatening event, followed by a period of maximum of 8 days to complete the initial preliminary report. All other SAEs will be reported within a period of maximum 15 days after sponsor has first knowledge of the serious adverse events.

7.3 Follow-up of adverse events All AEs will be followed until they have abated, or until a stable situation has been reached. Depending on event, follow up may require additional tests or medical procedures as indicated, and/or referral to general physician or medical specialist. SAEs need to be reported till end of study (last follow up moment for last subject), as defined in the protocol.

8. STATISTICAL ANALYSIS 8.1 Primary study parameter(s) The primary study parameter is to define if the normal sequence of segmental contributions in the lower cervical spine during the second half of extension (C4-C5 followed by C5-C6, and then C6-C7) is present in asymptomatic participants between 55 and 70 years of age by using cinematographic recordings. Participants are seated on a crutch, adjustable in height, with their neck, shoulders and head free. As soon as the recording is started, the participant is instructed to move his head in the sagittal plane from maximal extension to maximal flexion, without moving the upper part of the body, in about 16 seconds. Participants perform this procedure twice with an interval of two weeks. Images will be analysed using computer software that uses an algorithm to follow motion of the vertebrae during complete flexion and extension. This will be done by two researchers for 4 cinematographic recordings to determine reproducibility using two way mixed, absolute agreement, intra-class correlation coefficient. Graphs will be made for flexion and extension in which segmental rotation between each pair of successive frames of each individual segment within C4 to C7 will be plotted against the cumulative rotation in segments C4 to C7 together (block C4-C7) to describe the sequence of segmental contributions during flexion and extension. These graphs will be made and analysed for each individual participant to determine if the normal sequence of segmental contributions is present or absent. T1 will be tested against T2 using coefficient of variation and intra-individual standard deviation to determine if the defined sequence is consistent between two recordings in the intra-individual variability.

8.2 Secondary study parameter(s) The secondary study parameter is defining the sROM of C4-C5, C5-C6 and C6- C7 by analysing the flexion and extension cinematographic recordings in asymptomatic participants between 55 and 70 years of age. Rotation within a segment is calculated between each pair of successive frames to be able to determine the sequence of segmental contributions. All these small rotations from extension to flexion (or vice versa) can be summated to calculate sROM for that motion segment.

9. ETHICAL CONSIDERATIONS 9.1 Regulation statement This research is conducted according to principles enshrined in the Declaration of Helsinki (3th edition 2013) and in accordance with the Medical Research Involving Human Subjects Act (WMO, version 1 July 2012).

9.2 Recruitment and consent Participants will be recruited from Zuyd Hogeschool Sittard/Heerlen and Zuyderland Medical Center Sittard-Geleen/Heerlen using posters. Possible participants have to contact the researcher by email if they are interested in participation. Further information will be given verbally and in writing, followed by a thinking time of seven days. When people are willing to participate and meet the inclusion criteria, informed consent will be signed during the first meeting between researcher and participant. Participants can terminate their participation at all times, without giving a reason. For any questions regarding the study, an independent physician is available throughout the duration of the study.

9.3 Objection by minors or incapacitated subjects (if applicable) Not applicable.

9.4 Benefits and risks assessment, group relatedness Participants do not directly benefit from participating in this study. They make a contribution to knowledge in the field of motion of the cervical spine in the elderly population. Increased knowledge of physiological motion enables us to recognize abnormal motion in future. Phantom measurements of the Alura Xper in Zuyderland Sittard were used to determine radiation dosage. According to radiation experts, radiation dosage per cinematographic recording will be 0.084 mSv. Participants will perform cinematographic recordings twice, resulting in a total radiation dose of 0.168 mSv. Moreover, before definitive inclusion in the study a lateral X-ray of the cervical spine will be performed to determine eligibility resulting in a radiation dose of 0.0096 mSv. Total radiation dose per participant will therefore be 0.1776 mSv. This amount of radiation can be categorized in category IIa using the NCS guidelines about risks of radiation dosage (0.1 to 1 mSv). This category includes moderate risk which can be justified if there is a potential health benefit for future patients.

9.5 Compensation for injury The sponsor/investigator has a liability insurance which is in accordance with article 7 of the WMO. The sponsor (also) has an insurance which is in accordance with the legal requirements in the Netherlands (Article 7 WMO). This insurance provides cover for damage to re- search subjects through injury or death caused by the study. The insurance applies to the damage that becomes apparent during the study or within 4 years after the end of the study.

9.6 Incentives (if applicable) Participants will be reimbursed for extra time that is needed to fill out the questionnaires and undergo cinematographic recordings. They will receive €50 for participating in T1 and T2. Participants that live outside of Sittard will receive mission expenses of €0.20 per kilometre.

10. ADMINISTRATIVE ASPECTS, MONITORING AND PUBLICATION 10.1 Handling and storage of data and documents Data will be stored in two ways; cinematographic recordings on CDs and questionnaires on paper. Both of them will be coded with participant-number (e.g. participant 5). Cinematographic recordings will also be coded with recording-number (e.g. recording 5). CDs and questionnaires will be locked up in a secured room in the Maastricht University Medical Centre (MUMC+). Data analysis will also take place in the MUMC+. Data will be kept for 15 years after ending the study. Handling of personal data will comply with the Dutch Personal Data Protection Act (Wbp).

10.2 Monitoring and Quality Assurance Monitoring will be performed by trained and qualified monitors. According to Good Clinical Practice (GCP) guidelines main task of the monitor is ensuring that: Rights and well-being of human participants are protected.

Reported trial data are accurate, complete and verifiable from source documents.

Conduct of trial is in compliance with currently approved protocol, GCP and applicable regulatory requirements.

Prior to the study start a monitoring plan will be assembled, specifying Source Document Verification Plan, frequency of monitoring visits and frequency of checking Trial Master Files/Investigator Site Files.

Monitoring will be performed remotely and on site.

There are several kinds of monitoring visits:

Site initiation visit (SIV): SIV will be performed after all approvals have been obtained and prior to enrolling the first subject in that centre.

Interim monitoring visit (IMV): Several IMV's will be performed during the trial.

Frequency of visits is determined in monitoring plan.

- Close out visit (COV): COV will be performed at the end of the trial, after collection of all data. Monitoring visits will be planned in agreement with study site personnel. According to GCP guidelines, the investigators must provide the monitor with all necessary information and documents. Furthermore, the investigators are obliged to answer all queries raised by monitor in eCRF in timely manner. After each monitoring visit, a follow-up email with all action points will be sent to the study site. These action points will be addressed at beginning of the next monitoring visit.

10.3 Amendments Amendments are changes made to the research after a favourable opinion by the accredited METC has been given. All amendments will be notified to the METC that gave a favourable opinion.

10.4 Annual progress report The researcher will submit a summary of progress of the trial to the accredited METC once a year. Information will be provided on date of inclusion of the first subject, numbers of subjects included and numbers of subjects that have completed the trial, serious adverse events, other problems, and amendments.

10.5 Temporary halt and (prematurely) end of study report The researcher will notify the accredited METC of the end of the study within a period of 8 weeks. The end of the study is defined as the last participants' last visit. The researcher will notify METC immediately of a temporary halt of the study, including reason of such an action. In case of ending the study prematurely, the researcher will notify the accredited METC within 10 days, including reasons for premature termination. Within one year after the end of the study, the researcher will submit a final study report with results, including any publications/abstracts, to the accredited METC.

10.6 Public disclosure and publication policy This trial will be registered in a public trial register before recruitment of the first participant. Results will preferable be published in open access, peer-reviewed journals. Data of participants will be anonymous for publication and cannot be traced to an individual. In case of negative results, data will also be published. Possible funding has through contractual agreement no effect on publication. There is no veto over whether or not to publish data by one of the parties.

ELIGIBILITY:
Inclusion Criteria:

1. Age 55-70 years.
2. Ability to actively perform flexion/extension movements of the neck without pain or other symptoms.
3. No history of neck complaints.
4. Neck Disability Index (NDI) score of 4 or less.
5. Kellgren's score of 3 or less.
6. Informed consent

Exclusion Criteria:

1. Previous surgery on the cervical spine.
2. Symptoms of cervical radiculopathy of myelopathy (e.g. positive Lhermitte's sign).
3. Active infection.
4. Immature bone.
5. Previous or actual tumorous processes in the cervical region.
6. Previous radiation therapy in the cervical region.
7. Not able to speak Dutch.

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Physiologic motion pattern of the lower cervical spine | Two recordings will be made with an interval of two weeks and will be analysed within one year. Change will not be assesed. Recordings are made in the same individual at two time points to have to independent objective measurements.
  The normal sequence of segmental contributions in the lower cervical spine (C4-C5 followed by C5-C6, and then C6-C7) during the second half of extension in asymptomatic participants

SECONDARY OUTCOMES:
Segmental ROM of C4-C5, C5-C6, and C6-C7 | Two recordings will be made with an interval of two weeks and will be analysed within one year. Change will not be assesed. Recordings are made in the same individual at two time points to have to independent objective measurements.
  Analysing the flexion and extension cinematographic recordings in asymptomatic participants

CONTACTS AND LOCATIONS:
Overall Officials: Henk Van Santbrink, MD, PhD, Prof, Principal Investigator — Maastricht University Medical Centre
Locations (1):
- Zuyderland Medisch Centrum, Heerlen, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The patient data (screening information and cinematographic recordings) will be made available to drs. Smeets and drs. Schuermans for analysis
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: The data will be available for the duration of the study, which is estimated to be one year. Data will be stored safely at the MUMC for 15 years.

REFERENCES:
- [Background] Bogduk N, Mercer S. Biomechanics of the cervical spine. I: Normal kinematics. Clin Biomech (Bristol). 2000 Nov;15(9):633-48. doi: 10.1016/s0268-0033(00)00034-6. PMID 10946096
- [Background] Van Mameren H, Drukker J, Sanches H, Beursgens J. Cervical spine motion in the sagittal plane (I) range of motion of actually performed movements, an X-ray cinematographic study. Eur J Morphol. 1990;28(1):47-68. PMID 2390411
- [Background] Boselie TFM, van Santbrink H, de Bie RA, van Mameren H. Pilot Study of Sequence of Segmental Contributions in the Lower Cervical Spine During Active Extension and Flexion: Healthy Controls Versus Cervical Degenerative Disc Disease Patients. Spine (Phila Pa 1976). 2017 Jun 1;42(11):E642-E647. doi: 10.1097/BRS.0000000000001914. PMID 27879563
- [Background] Reinartz R, Platel B, Boselie T, van Mameren H, van Santbrink H, Romeny Bt. Cervical vertebrae tracking in video-fluoroscopy using the normalized gradient field. Med Image Comput Comput Assist Interv. 2009;12(Pt 1):524-31. doi: 10.1007/978-3-642-04268-3_65. PMID 20426028
- [Background] Simpson AK, Biswas D, Emerson JW, Lawrence BD, Grauer JN. Quantifying the effects of age, gender, degeneration, and adjacent level degeneration on cervical spine range of motion using multivariate analyses. Spine (Phila Pa 1976). 2008 Jan 15;33(2):183-6. doi: 10.1097/BRS.0b013e31816044e8. PMID 18197104
- [Background] Lansade C, Laporte S, Thoreux P, Rousseau MA, Skalli W, Lavaste F. Three-dimensional analysis of the cervical spine kinematics: effect of age and gender in healthy subjects. Spine (Phila Pa 1976). 2009 Dec 15;34(26):2900-6. doi: 10.1097/BRS.0b013e3181b4f667. PMID 20010397
- [Background] Cote P, Cassidy JD, Yong-Hing K, Sibley J, Loewy J. Apophysial joint degeneration, disc degeneration, and sagittal curve of the cervical spine. Can they be measured reliably on radiographs? Spine (Phila Pa 1976). 1997 Apr 15;22(8):859-64. doi: 10.1097/00007632-199704150-00007. PMID 9127918
- [Background] Boselie TF, van Mameren H, de Bie RA, van Santbrink H. Cervical spine kinematics after anterior cervical discectomy with or without implantation of a mobile cervical disc prosthesis; an RCT. BMC Musculoskelet Disord. 2015 Feb 21;16:34. doi: 10.1186/s12891-015-0479-4. PMID 25887569
- [Background] KELLGREN JH, LAWRENCE JS. Radiological assessment of osteo-arthrosis. Ann Rheum Dis. 1957 Dec;16(4):494-502. doi: 10.1136/ard.16.4.494. No abstract available. PMID 13498604
- [Background] Vernon H, Mior S. The Neck Disability Index: a study of reliability and validity. J Manipulative Physiol Ther. 1991 Sep;14(7):409-15. PMID 1834753
- [Derived] Schuermans VNE, Smeets AYJM, Breen A, Branney J, Curfs I, van Santbrink H, Boselie TFM. An observational study of quality of motion in the aging cervical spine: sequence of segmental contributions in dynamic fluoroscopy recordings. BMC Musculoskelet Disord. 2024 Apr 25;25(1):330. doi: 10.1186/s12891-024-07423-z. PMID 38664811
- See also: Related Info — https://radiationdosimetry.org/ncs/documents/ncs-26-human-exposure-to-ionising-radiation-for-clinical-and-research-purposes-radiation-dose-risk-estimates